CLINICAL TRIAL: NCT00731094
Title: Expert System-Based Feedback in Sedentary Overweight Veterans
Brief Title: The VA-STRIDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Brown University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 07-154
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obesity; Sedentary Lifestyle
Keywords: overweight; sedentary lifestyle; exercise; primary health care; controlled clinical trials, randomized
MeSH Terms: conditions — Overweight; Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): Expert system-based physical activity counseling: Individualized baseline counseling and guided goal setting to increase physical activity gradually to at least 150 minutes/week of moderate intensity, with a 12-month follow-up via postal mail of 14 additional counseling contacts generated by responses to a physical activity questionnaire and individually tailored computer-generated expert system feedback messages for physical activity based on stages of the motivational readiness for change model
  Interventions: Behavioral: Expert system-based physical activity counseling
- Attention Control (No Intervention): Generalized baseline healthy lifestyle education and suggestion to increase physical activity, with a 12-month follow-up via postal mail of 14 wellness newsletters focused on health issues other than physical activity

INTERVENTIONS:
Behavioral: Expert system-based physical activity counseling — The intervention included 14 mailings to participants that involved completion of physical activity questionnaires printed on forms that were scanned into a computerized expert system program to generate individually-tailored feedback messages and related manuals based on the Stages of Motivational Readiness for Change Model. Newsletters providing additional support and suggestions for increasing physical activity were also part of the mailing program.
  Arms: Physical Activity Intervention

SUMMARY:
The purpose of the study was to examine the effectiveness of an expert-system, print-based physical activity (PA) intervention delivered to Veterans receiving primary care at the VA Pittsburgh Healthcare System (VAPHS).

DETAILED DESCRIPTION:
A.1 The primary aim of the study was to determine the effect of a physical activity intervention designed to increase physical activity for sedentary Veterans at VAPHS.

A.2. Secondary aims were to assess key health-related outcomes related to the intervention including health and quality of life. The specific outcomes were to (a) estimate the impact of the intervention on physical function, health-related quality of life (HRQL), weight, blood pressure, and serum lipids; and (b) characterize variation in intervention effectiveness by participant sociodemographic and health characteristics, such as age, race, and baseline health status.

232 Veterans were randomized to either the physical activity intervention group or the attention control group. Participants randomized to the physical activity intervention group participated in an individualized physical activity counseling session at baseline, conducted by an exercise physiologist, with guided goal setting to increase physical activity gradually to at least 150 minutes/week of moderate intensity. An additional 14 intervention counseling contacts, generated by participants' responses to physical activity questionnaires and individually tailored computer-generated expert system feedback messages based on stages of the motivational readiness for change model, were conducted via postal mail over the subsequent 12 months in parallel with routine primary care. Newsletters providing additional support and suggestions for increasing physical activity were also part of the mailed counseling contacts. Participants randomized to the attention control group participated in a generalized healthy lifestyle counseling session at baseline, conducted by a health educator, which included limited advice to become more physically active. Fourteen follow-up wellness newsletters that focused on healthy lifestyle issues other than physical activity were sent to participants via postal mail over the subsequent 12 months with the same frequency of contact as for the physical activity intervention group and in parallel with routine primary care. Assessment of effectiveness occurred at baseline, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age at the time of enrollment,
* one or more primary care clinic visits at VAPHS in the 12 months prior to enrollment
* overweight or obese, with a BMI > =25.0 kg/m^2 at the most recent primary care visit prior to enrollment.

Exclusion Criteria:

* primary care provider judgment that unsupervised moderate-intensity exercise will place the Veteran at risk of a cardiovascular event, or other safety concern for guided but unsupervised physical activity
* Veteran is nonambulatory or requires assistive devices to ambulate (e.g., wheelchairs, prosthetic legs, canes or walkers),
* Veteran regularly participates in moderate to brisk physical activity 60 minutes or more each week
* current diagnosis of pulmonary hypertension, chronic obstructive pulmonary disease (COPD), and other comorbid conditions deemed to be contraindications for guided, unsupervised physical activity
* self-reported blindness and/or unable to read printed material in English (e.g., a newspaper)
* plans to move from the VAPHS treatment area in the next 12 months
* unable or unwilling to travel to the study site 4 times during the 12-month study period
* VAPHS employee
* current participant in another interventional research study that may confound outcomes
* unable or unwilling to provide signed, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Sevick, ScD MS, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Hawkins MS, Hough LJ, Berger MA, Mor MK, Steenkiste AR, Gao S, Stone RA, Burkitt KH, Marcus BH, Ciccolo JT, Kriska AM, Klinvex DT, Sevick MA. Recruitment of veterans from primary care into a physical activity randomized controlled trial: the experience of the VA-STRIDE study. Trials. 2014 Jan 7;15:11. doi: 10.1186/1745-6215-15-11. PMID 24398076
- [Derived] Gao S, Stone RA, Hough LJ, Haibach JP, Marcus BH, Ciccolo JT, Kriska AM, Burkitt KH, Steenkiste AR, Berger MA, Sevick MA. Physical activity counseling in overweight and obese primary care patients: Outcomes of the VA-STRIDE randomized controlled trial. Prev Med Rep. 2015 Dec 21;3:113-20. doi: 10.1016/j.pmedr.2015.12.007. eCollection 2016 Jun. PMID 26844197

RESULTS

PARTICIPANT FLOW:
Groups:
- Physcial Activity Intervention: Individualized baseline counseling and guided goal setting to increase physical activity gradually to at least 150 minutes/week of moderate intensity, with a 12-month follow-up via postal mail of 14 additional counseling contacts generated by responses to a physical activity questionnaire and individually tailored computer-generated expert system feedback messages for physical activity based on stages of the motivational readiness for change model
Period: Overall Study
Arm/Group | Physcial Activity Intervention | Attention Control
Started | 116 | 116
Month 6 | 101 | 107
Completed | 98 | 105
Not Completed | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physcial Activity Intervention | Attention Control | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (12.5) | 62.6 (13.2) | 63.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 96 | 96 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 111 | 113 | 224
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 26 | 54
  White | 86 | 87 | 173
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 116 | 116 | 232
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.1 (4.7) | 32.2 (5.0) | 31.6 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Moderate Intensity Physical Activity: Modified Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire
Description: Participants achieving 150 minutes/week of moderate intensity or greater physical activity at Month 0 as measured with the modified CHAMPS Questionnaire
Time Frame: Month 0
Measure: Number; unit: participants
Groups:
- Physical Activity Intervention: Individualized baseline counseling and guided goal setting to increase physical activity gradually to at least 150 minutes/week of moderate intensity, with a 12-month follow-up via postal mail of 14 additional counseling contacts generated by responses to a physical activity questionnaire and individually tailored computer-generated expert system feedback messages for physical activity based on stages of the motivational readiness for change model
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 116 | 116
participants | 37 | 44

2. Primary Outcome: Moderate Intensity Physical Activity: Modified CHAMPS Questionnaire
Description: Participants achieving 150 minutes/week of moderate intensity or greater physical activity at Month 6 as measured with the modified CHAMPS Questionnaire
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 101 | 106
participants | 48 | 53

3. Primary Outcome: Moderate Intensity Physical Activity: Modified CHAMPS Questionnaire
Description: Participants achieving 150 minutes/week of moderate intensity or greater physical activity at Month 12 as measured with the modified CHAMPS Questionnaire
Time Frame: Month 12
Measure: Number; unit: participants
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 97 | 105
participants | 52 | 49

4. Primary Outcome: Moderate Intensity Physical Activity: Accelerometer
Description: Participants with an average of at least 30 minutes/day of moderate intensity or greater physical activity in a subset of the study population for whom accelerometer data were obtained: 97 of 116 in Physical Activity Intervention Group and 103 of 116 in Attention Control Group at Month 0
Time Frame: Month 0
Measure: Number; unit: participants
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 97 | 103
participants | 31 | 36

5. Primary Outcome: Moderate Intensity Physical Activity: Accelerometer
Description: Participants with an average of at least 30 minutes/day of moderate intensity or greater physical activity in a subset of the study population for whom accelerometer data were obtained: 77 of 101 in Physical Activity Intervention Group and 76 of 107 in Attention Control Group in Month 6
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 77 | 76
participants | 26 | 19

6. Primary Outcome: Moderate Intensity Physical Activity: Accelerometer
Description: Participants with an average of at least 30 minutes/day of moderate intensity or greater physical activity in a subset of the study population for whom accelerometer data were obtained: 71 of 98 in Physical Activity Intervention Group and 74 of 105 in Attention Control Group at Month 12
Time Frame: Month 12
Measure: Number; unit: participants
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 71 | 74
participants | 24 | 21

7. Secondary Outcome: Weight
Description: Weight in kilograms (kg) measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 116 | 116
kg | 95.5 (16.9) | 98.7 (17.3)

8. Secondary Outcome: Weight
Description: Weight in kilograms at measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 101 | 106
kg | 95.2 (17.5) | 97.7 (17.7)

9. Secondary Outcome: Weight
Description: Weight in kilograms measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 98 | 104
kg | 95.3 (17.5) | 98.0 (17.4)

10. Secondary Outcome: Systolic Blood Pressure (BP)
Description: Systolic BP in millimeters of mercury (mmHg) measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 116 | 116
mmHg | 126.1 (17.8) | 126.1 (14.2)

11. Secondary Outcome: Systolic BP
Description: Systolic BP measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 97 | 104
mmHg | 129.1 (17.8) | 130.1 (16.0)

12. Secondary Outcome: Systolic BP
Description: Systolic BP measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 98 | 101
mmHg | 130.0 (18.3) | 129.3 (16.9)

13. Secondary Outcome: Diastolic BP
Description: Diastolic BP measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 116 | 116
mmHg | 73.1 (9.7) | 74.1 (9.5)

14. Secondary Outcome: Diastolic BP
Description: Diastolic BP measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 97 | 104
mmHg | 73.7 (10.8) | 75.7 (10.0)

15. Secondary Outcome: Diastolic BP
Description: Diastolic BP measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 98 | 101
mmHg | 74.4 (10.3) | 75.9 (9.9)

16. Secondary Outcome: Low-density Lipoprotein (LDL) Cholesterol
Description: LDL cholesterol in milligrams per deciliter (mg/dL) measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 95 | 108
mg/dL | 95.3 (33.7) | 96.4 (33.1)

17. Secondary Outcome: LDL Cholesterol
Description: LDL cholesterol measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 77 | 75
mg/dL | 91.6 (33.4) | 95.8 (29.3)

18. Secondary Outcome: LDL Cholesterol
Description: LDL cholesterol measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 49 | 50
mg/dL | 92.4 (31.9) | 96.8 (39.2)

19. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol
Description: HDL cholesterol in milligrams/deciliter (mg/dL) measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 95 | 108
mg/dL | 45.4 (12.6) | 43.2 (11.1)

20. Secondary Outcome: HDL Cholesterol
Description: HDL cholesterol measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 77 | 75
mg/dL | 46.0 (12.9) | 44.4 (10.2)

21. Secondary Outcome: HDL Cholesterol
Description: HDL cholesterol measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 49 | 50
mg/dL | 45.8 (13.4) | 44.3 (11.3)

22. Secondary Outcome: Triglycerides
Description: Triglycerides measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 95 | 105
mg/dL | 132.9 (73.6) | 134.4 (87.4)

23. Secondary Outcome: Triglycerides
Description: Triglycerides measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 77 | 75
mg/dL | 128.5 (73.5) | 139.7 (88.1)

24. Secondary Outcome: Triglycerides
Description: Triglycerides measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 49 | 50
mg/dL | 145.8 (81.8) | 144.2 (95.4)

25. Secondary Outcome: Health Related Quality of Life (HRQL): Short Form 36 Health Survey Questionnaire (SF-36) Physical Component Summary Measure (PCS)
Description: HRQL: SF-36 PCS measured at Month 0. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The PCS aggregates the scales for bodily pain, general health perceptions, physical functioning, and role limitation due to physical health problems.
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 115 | 116
scores on a scale | 44.7 (8.3) | 47.0 (8.3)

26. Secondary Outcome: HRQL: SF-36 PCS
Description: HRQL: SF-36 PCS measured at Month 6. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The PCS aggregates the scales for bodily pain, general health perceptions, physical functioning, and role limitation due to physical health problems.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 101 | 106
scores on a scale | 45.4 (8.1) | 45.4 (8.9)

27. Secondary Outcome: HRQL: SF-36 PCS
Description: HRQL: SF-36 PCS measured at Month 12. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The PCS aggregates the scales for bodily pain, general health perceptions, physical functioning, and role limitation due to physical health problems.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 98 | 104
scores on a scale | 44.9 (9.3) | 45.1 (9.5)

28. Secondary Outcome: HRQL: SF-36 Mental Component Summary Measure (MSC)
Description: HRQL: SF-36 MCS measured at Month 0. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The MCS aggregates the scales for vitality, mental health, social functioning, and role limitations due to personal or emotional problems.
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 115 | 116
scores on a scale | 51.6 (9.6) | 53.0 (8.6)

29. Secondary Outcome: HRQL: SF-36 MCS
Description: HRQL: SF-36 MCS measured at Month 6. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The MCS aggregates the scales for vitality, mental health, social functioning, and role limitations due to personal or emotional problems.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 101 | 107
scores on a scale | 51.3 (10.8) | 51.6 (9.4)

30. Secondary Outcome: HRQL: SF-36 MCS
Description: HRQL: SF-36 MCS measured at Month 12. The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The 8 scales are the weighted sums of the 2-10 questions in their section. Norm-based scoring, where each scale and component summary measures were scored to have the same average (50) and the same standard deviation (10 points), was used for reporting results in this study. Scores are interpreted as the lower the score the more disability; conversely, the higher the score the less disability. The MCS aggregates the scales for vitality, mental health, social functioning, and role limitations due to personal or emotional problems.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 98 | 104
scores on a scale | 53.0 (9.5) | 52.8 (8.4)

31. Secondary Outcome: Physical Function: 6-Minute Walking Distance (6MWD)
Description: Physical Function: 6MWD in meters measured at Month 0
Time Frame: Month 0
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 115 | 115
meters | 435.9 (88.7) | 445.5 (100.3)

32. Secondary Outcome: Physical Function: 6MWD
Description: Physical Function: 6MWD measured at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 87 | 92
meters | 453.9 (79.8) | 458.5 (105.9)

33. Secondary Outcome: Physical Function: 6MWD
Description: Physical Function: 6MWD measured at Month 12
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Activity Intervention | Attention Control
Number analyzed (Participants) | 88 | 85
meters | 457.5 (81.4) | 444.9 (127.2)

ADVERSE EVENTS:
Time Frame: Data for adverse events were collected during the 12-month follow-up period.
Description: The systematic assessment for adverse events was conducted via monthly telephone interviews with enrolled participants.
Arm/Group | Physical Activity Intervention | Attention Control
Serious Adverse Events (participants affected / at risk) | 29/116 | 33/116
Other Adverse Events (participants affected / at risk) | 0/116 | 0/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Physical Activity Intervention (N=116) | Attention Control (N=116)
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac catheterization (Cardiac disorders) | 1 | 2
Chest pains/pressure (Cardiac disorders) | 2 | 6
Acid reflux/vomiting (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Gallbladder problems (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Eye trauma (Injury, poisoning and procedural complications) | 1 | 1
Sleep apnea (Investigations) | 2 | 3
Vertigo (Investigations) | 1 | 1
Nerve pain (Nervous system disorders) | 1 | 0
Anxiety/stress (Psychiatric disorders) | 0 | 1
Kidney stones (Renal and urinary disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Fluid retention in leg (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract surgery (Surgical and medical procedures) | 3 | 2
Colectomy (Surgical and medical procedures) | 1 | 0
Hernia surgery (Surgical and medical procedures) | 0 | 2
Knee/ankle surgery (Surgical and medical procedures) | 0 | 2
Lymphadenectomy (Surgical and medical procedures) | 1 | 0
Pacemaker inserted (Surgical and medical procedures) | 1 | 1
Prostate surgery (Surgical and medical procedures) | 0 | 1
Shoulder surgery (Surgical and medical procedures) | 2 | 0
Transient ischemic attack (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No